CLINICAL TRIAL: NCT05501522
Title: A Phase III, Placebo-controlled, Randomized, Observer-blinded, Multi-national, Multi-center Study to Assess the Safety, Reactogenicity, and Immunogenicity of Heterologous Booster Vaccination of a SARS-CoV-2 Recombinant Protein Nanoparticle Vaccine (GBP510) Adjuvanted with AS03 in Adults Aged 18 Years and Older
Brief Title: Immunogenicity and Safety Study of Heterologous Booster Vaccination of a SARS-CoV-2 Recombinant Protein Nanoparticle Vaccine(GBP510) Adjuvanted with AS03 in Adults Aged 18 Years and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Bioscience Co., Ltd. (Industry)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other); International Vaccine Institute (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GBP510_004
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — GBP510 vaccine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (12):
- Primary series of mRNA-1273 manufactured by ModernaTX, Inc. (Experimental): participants who received primary vaccination of a mRNA-1273 at least 12 weeks prior to study vaccination will be enrolled and block-randomized in 6:1 ratio to receive one dose of GBP510 adjuvanted with AS03 (Test Vaccine).
  Interventions: Biological: GBP510 adjuvanted with AS03
- Primary series of mRNA-1273 manufactured by ModernaTX, Inc. (Placebo) (Placebo Comparator): participants who received primary vaccination of a mRNA-1273 at least 12 weeks prior to study vaccination will be enrolled and block-randomized in 6:1 ratio to receive placebo.
  Interventions: Other: Placebo (Normal Saline)
- Primary series of ChAdOx1 nCOV-19 manufactured by Astrazeneca or S.I of India Pvt., Ltd. (Experimental): participants who received primary vaccination of a ChAdOx1 at least 12 weeks prior to study vaccination will be enrolled and block-randomized in 6:1 ratio to receive one dose of GBP510 adjuvanted with AS03 (Test Vaccine).
  Interventions: Biological: GBP510 adjuvanted with AS03
- Primary series of ChAdOx1 nCOV-19 manufactured by Astrazeneca or S.I of India Pvt., Ltd. (Placebo) (Placebo Comparator): participants who received primary vaccination of a ChAdOx1 at least 12 weeks prior to study vaccination will be enrolled and block-randomized in 6:1 ratio to receive placebo.
  Interventions: Other: Placebo (Normal Saline)
- A single dose vaccination of Ad26.COV2.S manufactured by Janssen Pharmaceuticals/Johnson & Johnson (Experimental): participants who received primary vaccination of a Ad26.COV2.S at least 12 weeks prior to study vaccination will be enrolled and block-randomized in 6:1 ratio to receive one dose of GBP510 adjuvanted with AS03 (Test Vaccine).
  Interventions: Biological: GBP510 adjuvanted with AS03
- A single dose vaccination of Ad26.COV2.S manufactured by Janssen Pharmaceuticals/J&J (Placebo) (Placebo Comparator): participants who received primary vaccination of a Ad26.COV2.S at least 12 weeks prior to study vaccination will be enrolled and block-randomized in 6:1 ratio to receive Placebo.
  Interventions: Other: Placebo (Normal Saline)
- Primary series of BNT162b2 manufactured by Pfizer/BioNTech (Active Comparator): participants who received primary vaccination of a BNT162b2 at least 12 weeks prior to study vaccination will be enrolled and block-randomized in 6:1 ratio to receive one dose of GBP510 adjuvanted with AS03 (Test Vaccine).
  Interventions: Biological: GBP510 adjuvanted with AS03
- Primary series of BNT162b2 manufactured by Pfizer/BioNTech (Placebo) (Placebo Comparator): participants who received primary vaccination of a BNT162b2 at least 12 weeks prior to study vaccination will be enrolled and block-randomized in 6:1 ratio to receive placebo.
  Interventions: Other: Placebo (Normal Saline)
- Primary series of BBIBP-CorV manufactured by Sinopharm (Experimental): participants who received primary vaccination of a BBIBP-CorV at least 12 weeks prior to study vaccination will be enrolled and block-randomized in 6:1 ratio to receive one dose of GBP510 adjuvanted with AS03 (Test Vaccine).
  Interventions: Biological: GBP510 adjuvanted with AS03
- Primary series of BBIBP-CorV manufactured by Sinopharm (Placebo) (Placebo Comparator): participants who received primary vaccination of a BBIBP-CorV at least 12 weeks prior to study vaccination will be enrolled and block-randomized in 6:1 ratio to receive placebo
  Interventions: Other: Placebo (Normal Saline)
- Primary series of CoronaVac (Active Comparator): participants who received primary vaccination of a CoronaVac at least 12 weeks prior to study vaccination will be enrolled and block-randomized in 6:1 ratio to receive one dose of GBP510 adjuvanted with AS03 (Test Vaccine).
  Interventions: Biological: GBP510 adjuvanted with AS03
- Primary series of CoronaVac (Placebo) (Placebo Comparator): participants who received primary vaccination of a CoronaVac at least 12 weeks prior to study vaccination will be enrolled and block-randomized in 6:1 ratio to receive one dose Placebo
  Interventions: Other: Placebo (Normal Saline)

INTERVENTIONS:
Biological: GBP510 adjuvanted with AS03 — injection volume of 0.5mL on Day 0
  Arms: A single dose vaccination of Ad26.COV2.S manufactured by Janssen Pharmaceuticals/Johnson & Johnson; Primary series of BBIBP-CorV manufactured by Sinopharm; Primary series of BNT162b2 manufactured by Pfizer/BioNTech; Primary series of ChAdOx1 nCOV-19 manufactured by Astrazeneca or S.I of India Pvt., Ltd.; Primary series of CoronaVac; Primary series of mRNA-1273 manufactured by ModernaTX, Inc.
Other: Placebo (Normal Saline) — injection volume of 0.5mL on Day 0
  Arms: A single dose vaccination of Ad26.COV2.S manufactured by Janssen Pharmaceuticals/J&J (Placebo); Primary series of BBIBP-CorV manufactured by Sinopharm (Placebo); Primary series of BNT162b2 manufactured by Pfizer/BioNTech (Placebo); Primary series of ChAdOx1 nCOV-19 manufactured by Astrazeneca or S.I of India Pvt., Ltd. (Placebo); Primary series of CoronaVac (Placebo); Primary series of mRNA-1273 manufactured by ModernaTX, Inc. (Placebo)

SUMMARY:
This is a Phase III, randomized, placebo-controlled, observer-blinded, parallel-group, multi-center study to assess the safety, reactogenicity, and immunogenicity of heterologous booster vaccination of SK SARS-CoV-2 recombinant protein nanoparticle vaccine (GBP510) adjuvanted with AS03 in adults aged 18 years and older.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety, reactogenicity, and immunogenicity of heterologous booster vaccination of a SARS-CoV-2 Recombinant Protein Nanoparticle Vaccine (GBP510) adjuvanted with AS03 in adults aged 18 years and older.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 years of age and older, at the time of signing the informed consent.
* Participants who are healthy or medically stable as determined by medical evaluation including medical history, physical examination, clinical laboratory tests, and medical judgement of the investigator.
* Participants who are able to attend all scheduled visits and comply with all study procedures.
* Participants who received primary vaccination of 1 of 6 different WHO EUA qualified COVID-19 vaccine (mRNA-1273, ChAdOx1 nCOV-19, Ad26.COV2.S, BNT162b2, BBIBP-CorV, CoronaVac) at least 12 weeks prior to study vaccination, and with no history of other COVID-19 vaccination, including booster doses.
* Participants who have a qualitative test result for antibody to SARS-CoV-2 nucleocapsid proteins at screening for assessment of previous SARS-CoV-2 infection
* Female participants of childbearing potential must agree to be heterosexually inactive, or agree to consistently use at least one acceptable method of contraception from at least 4 weeks prior to the study vaccination to 12 weeks after the study vaccination
* Female participants with a negative urine or serum pregnancy test at screening.
* Capable of giving signed informed consent as described in Appendix 10.1.3 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Any clinically significant respiratory symptoms (e.g. cough, sore throat), febrile illness (tympanic temperature >38°C), or acute illness within 72 hours prior to the study vaccination. A prospective participant should not be included until 72 hours after the condition has resolved.
* Concurrent or past SARS-CoV-2 infection within 12 weeks prior to the study vaccination confirmed by virological or serological testing
* History of virologically or serologically confirmed SARS, or MERS disease
* History of congenital, hereditary, acquired immunodeficiency, or autoimmune disease.
* History of bleeding disorder or thrombocytopenia which is contraindicating intramuscular vaccination in the investigator's opinion.
* History of hypersensitivity and severe allergic reaction (e.g. anaphylaxis, Guillain-Barre syndrome) to any vaccines or components of the study intervention.
* History of malignancy within 1 year prior to the study vaccination (with the exception of malignancy with minimal risk of recurrence at the discretion of the investigator).
* Significant unstable chronic or acute illness that, in the opinion of the investigator, might pose a health risk to the participant if enrolled, or could interfere with the protocol-specified activities, or interpretation of study results.
* Any other conditions which, in the opinion of the investigator, might interfere with the evaluation of the study objectives (e.g., alcohol or drug abuse, neurologic or psychiatric conditions).
* Female participants who are pregnant or breastfeeding.
* Receipt of any medications or vaccinations intended to prevent COVID-19 except for the pre-defined COVID-19 vaccines expected to be given prior to screening (mRNA-1273, ChAdOx1 nCOV-19, Ad26.COV2.S, BNT162b2, BBIBP-CorV, CoronaVac).
* Receipt of any vaccine within 4 weeks prior to the study vaccination or planned receipt of any vaccine from enrollment through 4 weeks after the study vaccination, except for influenza vaccination, which may be received at least 2 weeks prior to the study vaccination.
* Receipt of immunoglobulins and/or any blood or blood products within 12 weeks prior to the study vaccination.
* Chronic use (more than 2 consecutive weeks) of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy; or long-term systemic corticosteroid therapy (≥10mg prednisone/day or equivalent for more than 2 consecutive weeks) within 12 weeks prior to the study vaccination. The use of topical and nasal glucocorticoids will be permitted.
* Participation in another clinical study and receipt of study intervention within 4 weeks prior to the study vaccination, or concurrent, planned participation in another clinical study with study intervention during the study period.
* Investigators, or study staff who are directly involved in the conduct of this study or supervised by the investigator, and their respective family members.
* Donation of ≥450mL of blood product within 4 weeks prior to screening, or planned donation of blood product during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2024-08-17 (Actual)

PRIMARY OUTCOMES:
GMFR (Geometric Mean Fold Rise) of neutralizing antibody to SARS-CoV-2 measured by wild-type virus neutralization assay from baseline(Visit 2) to2 weeks post heterologous booster vaccinationfor each cohort | 2 weeks post heterologous booster vaccination for eachcohort
  For all cohort

SECONDARY OUTCOMES:
GMT of neutralizing antibody to SARS-CoV-2 measured by wild-type virus neutralization assay at each time point post heterologous booster vaccination. | Through Day 365 post vaccination
  For all cohort
GMFR of neutralizing antibody to SARS-CoV-2 measured by wild-type virus neutralization assay from baseline (Visit 2) to each subsequent time point post heterologous booster vaccination. | Through Day 365 post vaccination
  For all cohort
Percentage of participants with ≥4-fold rise in wild-type virus neutralizing antibody titer to SARS-CoV-2 from baseline (Visit 2) to each subsequent time point post heterologous booster vaccination. | Through Day 365 post vaccination
  For all cohort
GMT of SARS-CoV-2 RBD-binding IgG antibody measured by ELISA at each time point post heterologous booster vaccination | Through Day 365 post vaccination
  For all cohort
GMFR of SARS-CoV-2 RBD-binding IgG antibody measured by ELISA from baseline (Visit 2) to each subsequent time point post heterologous booster vaccination | Through Day 365 post vaccination
  For all cohort
Percentage of participants with ≥4-fold rise in ELISA SARS-CoV-2 RBD-binding IgG titer from baseline (Visit 2) to each subsequent time point post heterologous booster vaccination. | Through Day 365 post vaccination
  For all cohort
Cell-mediated response for both Th1 and Th2 cytokines measured by ELISpot and/or FluoroSpot, and for both CD4+ and CD8+ T-cells measured by FACS | Through Day 365 post vaccination
  For all cohort (in a subset of participants)
Occurrence of immediate systemic reactions in 30 minutes post heterologous booster vaccination. | Through 30 minutes post booster vaccination
  For all cohort
Occurrence of solicited local/systemic Adverse Events(AEs) | Through 7 days post booster vaccination
  For all cohort
Occurrence of unsolicited AEs | Through 28 days post booster vaccination
  For all cohort
Occurrence of SAEs, MAAEs, AEs leading to study withdrawal, and AESIs during the whole study period. | Through Day 365 post booster vaccination
  Through 7 days post booster vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Santa K Das, MD, Principal Investigator — Institute of Medicine (IOM).
Locations (4):
- Colombia (2):
  - Policlínico Social Del Norte, Bogotá, Bogota D.C.
  - CAIMED (Centro de Atención e Investigación Médica), Chía, Cundinamarca
- Nepal (2):
  - Dhulikhel, Kathmandu, Dhulikhel
  - Institute of Medicine (IOM), Kathmandu, Maharajgunj

IPD SHARING:
Plan to Share IPD: No